CLINICAL TRIAL: NCT01884506
Title: Evaluation of the Effect of Body Weight and Composition on Iron Absorption and Blood Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Wageningen University (Other); Universidad de Monterrey (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof. Dr., Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: KEKZH-2013-0110
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- labeled iron meal (Experimental): Test meal (bread with honey) with a labeled iron solution
  Interventions: Dietary Supplement: labeled iron solution; Dietary Supplement: labeled iron solution and ascorbic acid
- labeled iron and ascorbic acid meal (Experimental): Test meal (bread with honey) with a labeled iron solution and ascorbic acid
  Interventions: Dietary Supplement: labeled iron solution; Dietary Supplement: labeled iron solution and ascorbic acid

INTERVENTIONS:
Dietary Supplement: labeled iron solution — labeled iron as ferrous sulfate (6mg/test meal)
Dietary Supplement: labeled iron solution and ascorbic acid — labeled iron as ferrous sulfate plus ascorbic acid (6mg:30mg /test meal)

SUMMARY:
A total of 75 subjects will be recruited for this study (25 normal weight, 25 overweight, 25 obese). In each subject blood volume will be determined using the minimally invasive carbon monoxide-rebreathing method (substudy 1) and iron absorption will be measured from a test meal labeled with stable iron isotopes. The effect of ascorbic acid on iron absorption will further be determined using a second labeled test meal (substudy 2). In addition, inflammation, hepcidin and iron status will be determined. In order to study the effect of body fat content on blood volume and iron absorption weight and height will be measured, and body fat will de determined by dual energy X-ray absorptiometry.

DETAILED DESCRIPTION:
Obesity has repeatedly been shown to be a risk factor for iron deficiency. The reason for this is believed to be reduced iron absorption as a result of increased circulating hepcidin concentrations. However, the direct interactions between body fat mass, iron absorption, inflammation and hepcidin have not been studied to date. Whether the low iron absorption in obese subjects could be overcome by conventional methods to increasing iron absorption, e.g. the addition of ascorbic acid and whether a reduction of inflammation could improve absorption is further unclear. For the calculation of fractional iron absorption from oral doses of stable iron isotopes an estimation of blood volume is required. Several equations to estimate blood volume from weight and height or calculated body surface area or volume are available, but have rarely been validated or used in obese subjects. The aim of the described study is therefore: 1) to determine blood volume using the carbon monoxide-rebreathing method over a large BMI range and to use those values to validate existing blood volume equations; 2) to measure iron absorption, hepcidin and inflammation in relation to BMI and body fat and 3) to assess the effect of ascorbic acid on iron absorption.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age 18-45 years
* Pre-menopausal (no absence of a menstrual cycle in the past 12 months)
* BMI 18.5-39.9 kg/m2 (n=25 18.5-24.9, n=25 25-29.9, n=25 30-39.9)
* Apparently healthy (no significant medical conditions that could influence iron or inflammatory status other than obesity (i.e., cancer, HIV/AIDS, inflammatory bowel disease, gastrointestinal bleeding, and rheumatoid arthritis, renal disease or hemochromatosis) (judged by study physician)

Exclusion Criteria:

* Moderate/sever anemia (Hb<11 g/dl)
* Use of medication which interferes with study measurements (judged by the study physician)
* Smoking
* Pregnancy and lactation; planning to become pregnant during the course of the study (pregnancy test will be conducted at visit 2 and subjects will be asked about contraception*)
* Consumption of vitamin- or mineral supplements unless they consent to discontinue intake two weeks before the start of the study until the final blood sampling
* Prior participation in studies using stable iron isotopes
* Food allergies/intolerances (gluten, lactose, milk protein)
* Blood donation during the two months prior to the study
* Major injuries during the 6 months prior to the study
* Illness during the 4 weeks prior to the study (judged by study physician)
* Administration of recombinant erythropoietin (rhEPO)
* More than 5 days at altitudes above 1600 m above sea level during the 3 weeks prior to the study
* Long distance flight (>8 h) during the 3 weeks prior to the study
* Chronic alcohol abuse

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption from the isotopically labeled test meals. | Baseline
  Iron absorption will be determined by incorporation of labeled iron into erythrocytes, 14 days after the administration of the last test meal containing labeled iron (stable isotope technique). Based on the shift of the iron isotope ratios in the blood samples and the amount of iron circulating in the body, the amounts of isotopic label iron present in the blood 14 days after the test meal administration will be calculated based on the principles of isotope dilution and considering that the iron isotopic labels are not monoisotopic. Circulating iron will be calculated based on blood volume as determined by carbon monoxide-rebreathing. For calculation of fractional absorption, 80% incorporation of the absorbed iron into red blood cells will be assumed.

SECONDARY OUTCOMES:
Hemoglobin mass will be measured with the carbon monoxide-rebreathing method. | Baseline
  Blood volume will be calculated from hemoglobin mass and compared to values determined by the different equations.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Aeberli, PhD, Principal Investigator — ETH Zurich
Locations (1):
- Human Nutrition Laboratory, ETH Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Cepeda-Lopez AC, Melse-Boonstra A, Zimmermann MB, Herter-Aeberli I. In overweight and obese women, dietary iron absorption is reduced and the enhancement of iron absorption by ascorbic acid is one-half that in normal-weight women. Am J Clin Nutr. 2015 Dec;102(6):1389-97. doi: 10.3945/ajcn.114.099218. Epub 2015 Nov 11. PMID 26561622